CLINICAL TRIAL: NCT02194816
Title: Modifiable Variables in Parkinsonism (MVP) [Formerly CAM Care in PD]
Brief Title: Modifiable Variables in Parkinsonism (MVP)
Status: Recruiting | Type: Observational
Sponsor: Bastyr University (Other)
Responsible Party: Principal Investigator, Laurie Mischley, Assistant Research Scientist, Bastyr University
Other Study IDs: BU-13A-1332
Record Dates: First submitted 2014-07-17; First posted 2014-07-18 (Estimated); Last update posted 2022-03-25 (Actual); Status verified 2022-03

CONDITIONS: Parkinson's Disease; Parkinsonism; MSA - Multiple System Atrophy; Progressive Supranuclear Palsy; Shy-Drager Syndrome; Corticobasal Degeneration; Dementia With Lewy Bodies; Pick Disease; Olivopontocerebellar Atrophies
Keywords: Parkinson's Disease; PD; Complementary and Alternative; CAM
MeSH Terms: conditions — Parkinson Disease; Parkinsonian Disorders; Shy-Drager Syndrome; Supranuclear Palsy, Progressive; Corticobasal Degeneration; Lewy Body Disease; Pick Disease of the Brain; Olivopontocerebellar Atrophies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Parkinson's Disease Patients: Any individuals who has a diagnosis of Parkinson's disease (PD), parkinsonism, or a parkinson's plus syndrome will be allowed to participate.

SUMMARY:
We are trying to identify factors associated with improved quality of life and fewer PD symptoms. We are attempting to identify practices, beliefs, and therapies used by individuals who report excellent quality of life, few PD symptoms, and reduced rates of progression. After agreeing to participate, we will ask participants to fill our questionnaires about their experience with PD, their health in general, along with their food intake every six months for five years.

DETAILED DESCRIPTION:
This is a prospective, observational study designed to describe disease progression, symptom change, quality of life, diet and lifestyle habits among patients with Parkinson's disease (PD). This study will identify and describe those individuals with the highest quality of life and least amount of disease activity, in order to describe medication, diet, and lifestyle patterns associated with a lack of PD disease progression and high quality of life.

Participants will be asked to complete online surveys every six months for five years. The time requirement is about an hour to an hour and a half every six months. Participants do not need to answer questions if they do not feel comfortable answering.

At each six month time point we will send participants an email with the link to the CAM Care in PD survey, a questionnaire about health and wellbeing (completed in REDCap). After participants have completed this survey we will send participants a link to the second survey, about dietary intake (completed on ASA24.gov). Because there is a designated window of time during which surveys must be completed, participants may receive a gentle reminder from us if time is running out.

This study is not designed to provide care. Participants are encouraged to consult with any providers you wish. Participants will not directly benefit from the study, but information gathered during the course of this study may help us begin to assess the longer-term effects of complementary and integrative care on health, disease progression and quality of life in PD patients.

ELIGIBILITY:
Inclusion Criteria:

* Parkinson's disease (PD)
* Parkinsonism
* Parkinson-plus syndromes (e.g. Multiple System Atrophy (MSA), Progressive Supranuclear Palsy (PSP), Corticobasal degeneration (CBGD), Dementia with Lewy bodies)
* Must have online access, an email address, basic computer literacy
* Must be willing to complete online surveys every 6 months for 5 years

Exclusion Criteria:

* Inability to read/write English
* Inability or unwillingness to complete surveys every six (6) months (~90 min)

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any individual with PD is invited to participate.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2012-09; Primary Completion 2030-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
CAM Care for PD survey | 5 years
  This survey has been developed to identify the complementary and alternative therapies most commonly used by individuals with PD. Results will be reported with descriptive statistics.
PROMIS: Global Health | 5 years
  This outcome measure will be used to assess general health and well-being in the cohort.
Patient-Reported Outcomes in PD (PRO-PD) | 5 years
  This outcome measure is a series of 33 slider bars, developed for this study, to evaluate the individual's perception of symptom severity. The cumulative score for all 33 listed symptoms will be reported as the PRO-PD score.

SECONDARY OUTCOMES:
Qualitative | 5 years
  Participants will be given 'free space' to provide additional information they consider relevant.

CONTACTS AND LOCATIONS:
Overall Officials: Laurie K Mischley, ND, PhD, MPH, Principal Investigator — Bastyr University
Locations (1):
- Bastyr University, Kenmore, Washington, United States

REFERENCES:
- [Background] Tomlinson CL, Stowe R, Patel S, Rick C, Gray R, Clarke CE. Systematic review of levodopa dose equivalency reporting in Parkinson's disease. Mov Disord. 2010 Nov 15;25(15):2649-53. doi: 10.1002/mds.23429. PMID 21069833
- [Background] Meissner WG, Frasier M, Gasser T, Goetz CG, Lozano A, Piccini P, Obeso JA, Rascol O, Schapira A, Voon V, Weiner DM, Tison F, Bezard E. Priorities in Parkinson's disease research. Nat Rev Drug Discov. 2011 May;10(5):377-93. doi: 10.1038/nrd3430. PMID 21532567
- [Background] Positive Deviance Initiative. 2010 [cited 2012 30 Dec 2012]; Available from: http://www.positivedeviance.org/about_pd/index.html